CLINICAL TRIAL: NCT02487823
Title: Phase Ib Dose Finding Study of BKM 120 in Combination With LH-RH Agonists and Bicalutamide in Men With Non Castrate Metastatic Prostate Cancer
Brief Title: Dose Finding Study of BKM 120 in Combination With LH-RH Agonists and Bicalutamide in Men With Non Castrate Metastatic Prostate Cancer
Acronym: NCMPC-BKM
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Defect of recruitment
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCMPC-BKM-IPC 2012-009
Record Dates: First submitted 2015-06-25; First posted 2015-07-02 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Non Castrate Metastatic Prostate Cancer
MeSH Terms: interventions — NVP-BKM120; Buserelin; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BKM 120 (60 mg) (Experimental): BKM120 (60 mg) in combination with LH-RH agonists and bicalutamide
  Interventions: Drug: BKM120 in combination with LH-RH agonists (suprefact) and bicalutamide
- BKM 120 (80 mg) (Experimental): BKM120 (80 mg) in combination with LH-RH agonists and bicalutamide
  Interventions: Drug: BKM120 in combination with LH-RH agonists (suprefact) and bicalutamide
- BKM 120 (100 mg) (Experimental): BKM120 (100 mg) in combination with LH-RH agonists and bicalutamide
  Interventions: Drug: BKM120 in combination with LH-RH agonists (suprefact) and bicalutamide

INTERVENTIONS:
Drug: BKM120 in combination with LH-RH agonists (suprefact) and bicalutamide — BKM 120, LH-RH agonists and Bicalutamide
  Other Names: BKM120, LH-RH agonists (suprefact) and bicalutamide (casodex)

SUMMARY:
To determine the maximum-tolerated dose (MTD) of BKM120 when administered orally in combination with daily bicalutamide and LH-RH agonists to men with non castrate metastatic prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer is the second leading cause of cancer and the third cause of death in male. Majority of patients had local disease that is cured by local treatment. Metastases are rare at the time of diagnosis but may occur after failure of local treatment (SEER).

Recommended treatment for non castrate metastatic prostate cancer (NCMPC) is castration by orchiectomy or medical castration by LH-RH (luteinizing hormone-releasing hormone) agonists alone and or combined androgen blockage with LH-RH agonists and anti androgen. Immediate treatment versus deferred treatment improve specific survival for advanced prostatic cancer : initial results of the Medical Research Council trial.

Continuous castration is superior to intermittent one with a median survival of 49 months. Chemotherapy combined with castration demonstrate a survival improvement compared to castration alone for high volume disease defined by visceral involvement and or 4 or more bone metastatis with almost one apendicular metastasis. For low volume disease or non selected metastatic hormone sensitive prostate cancer, Docetaxel demonstrated no survival benefit evaluated in a recent phase III trial (Sweeney C et al abs ASCO 2014).

However, most patients showing an initial response to hormonal therapy for advanced prostate cancer will progress to a castration-resistant phase of the disease with a much poorer prognosis. Median duration to androgen deprivation is 24 to 36 months, after patients become castrate resistant and docetaxel and other hormonal therapy like abiraterone and enzalutamide demonstrate survival improvement in castrate resistant prostate cancer.

Despite the considerable progress made with new agents such as abiraterone acetate or MDV3100 in metastatic castration resistant prostate cancer (mCRPC), new therapies are critical to improve castration sensitivity.

Understanding the mechanisms of resistance to AR and identifying directed new therapies is a real challenge in this situation.

Prostate cancer is characterized by its dependence on AR and its frequent activation of the Phosphatidylinositol-3-kinase (PI3K) pathway. Besides the resistance mediated by the mutation in the AR, among the non-steroid alternative pathways two major pathways have been associated with AR activation and CRPC, namely Ras/Raf/MEK/ERK and PI3K/AKT. More specifically a genomic profiling of human prostate cancer was recently reported where 42% of primary and 100% of the metastatic lesions studied had upregulated PI3K signaling mostly via loss of phosphatase activity such as PTEN (Phosphatase and tensin homolog) or INPP4B (inositol polyphosphate 4-phosphatase type II).

Dysregulation of the PI3K/PTEN pathway has also been associated with resistance to conventional antiandrogen therapies. Preclinical data support the potential for a reciprocal negative feedback between the AR and PI3K pathway.

Development of castration resistance is multifactorel including weak antagonist binding affi nity to AR, up-regulation of AR co-stimulatory pathways and increased intratumoural androgen levels as a result of intracrine androgen, as well as partial agonists properties of antiandrogens when AR is overexpressed.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (ICF) prior to screening
* Male patients (≥ 18 years)
* WHO performance status ≤ 2
* Histologically-confirmed adenocarcinoma of the prostate
* Patients with non castrate metastatic prostate cancer, with radiological metastatic disease ; patients with metastatic disease is documented on a Pet-Scan to choline is also eligible
* No previous chemotherapy treatment during the metastatic disease
* Neoadjuvant or adjuvant androgen deprivation therapy (ADT) treatment or for rising PSA is permitted if the ADT have been stopped for at least one year without metastasis or PSA increase during this time
* LH-RH agonists and bicalutamide had to began ≥ 28 days before registration
* Minimum pre treatment PSA > 5 ng/ml
* Patient has adequate bone marrow and organ function as defined by the following laboratory values:

  * Absolute Neutrophil Count (ANC) ≥ 1.0 x 109/L
  * Platelets ≥ 100 x 109/L
  * Hemoglobin ≥ 9.0 g/dL
  * INR ≤ 2
  * Potassium, calcium, magnesium within normal limits for the institution
  * Serum Creatinine ≤ 1.5 x ULN
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within normal range (or ≤ 3.0 x ULN if liver metastases are present)
  * Serum bilirubin within normal range (or ≤ 1.5 x ULN if liver metastases are present; or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert Syndrome)
  * Fasting plasma glucose (FPG) ≤ 120 mg/dL or ≤ 6.7 mmol/L 11. Agree to use effective contraception during the study and for at least 16 weeks after discontinuation 12. Patient is able to swallow and retain oral medication

Exclusion Criteria:

* Patients eligible for this study must not meet any of the following criteria:
* Patient has received previous treatment with PI3K and/or mTOR inhibitors
* Patient has a concurrent malignancy or has a malignancy within 3 years of study enrollment, (with the exception of adequately treated basal or squamous cell carcinoma or non-melanomatous skin cancer)
* ADT > 3 months
* Patient has any of the following mood disorders as judged by the Investigator or a Psychiatrist, or meets the cut-off score of ≥ 12 in the PHQ-9 or a cut-off of ≥ 15 in the GAD-7 mood scale, respectively, or selects a positive response of '1, 2, or 3' to question number 9 regarding potential for suicidal thoughts ideation in the PHQ-9 (independent of the total score of the PHQ-9):

  * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others) or patients with active severe personality disorders (defined according to DSM-IV) are not eligible Note: for patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous 6 weeks prior to start of study drug
  * ≥ CTCAE grade 3 anxiety
* Patient is concurrently using other approved or investigational antineoplastic agent Patient has received pelvic and/or para-aortic radiotherapy ≤ 28 days prior to enrollment in this study or has not recovered from side effects of such therapy at the time of initiation of screening procedures Patient has had major surgery within 28 days prior to starting study drug or has not recovered from major side effects of the surgery Patient has poorly controlled diabetes mellitus (HbA1c > 8 %) Patient with uncontrolled hypertension

Patient has active cardiac disease including any of the following:

* Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
* QTc > 480 msec on screening ECG (using the QTcF formula
* Angina pectoris that requires the use of anti-anginal medication
* Ventricular arrhythmias except for benign premature ventricular contractions
* Supraventricular and nodal arrythmias requiring a pacemaker or not controlled with medication
* Conduction abnormality requiring a pacemaker
* Valvular disease with documented compromise in cardiac function
* Symptomatic pericarditis

  - Patient has a history of cardiac dysfunction including any of the following:
* Myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
* History of documented congestive heart failure (New York Heart Association functional classification III-IV)
* Documented cardiomyopathy

  * Patient is currently receiving treatment with QT prolonging medication known to have a risk to induce Torsades de Pointes, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug
  * Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
  * Patient receiving chronic treatment with steroids or another immunosuppressive agent Note: Topical applications (e.g., rash), inhaled sprays (e.g., obstructive airways diseases), eye drops or local injections (e.g., intra-articular) are allowed. Patients with previously treated brain metastases, who are on a stable low dose corticosteroids treatment (e.g., dexamethasone 2 mg/day, prednisolone 10 mg/day) for at least 14 days before start of study treatment, are eligible
  * Patient has other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment contraindicate her participation in the clinical study (e.g.,chronic pancreatitis, active chronic hepatitis etc.)
  * Patient has a history of non-compliance to medical regimen
  * Patient is currently being treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug. Please refer to annex 9 for a list of prohibited CYP3A inhibitors and inducers Note: the oral anti-diabetic drugs troglitazone and pioglitazone are CYP3A inducers
  * Patient has a known history of HIV (testing not mandatory) infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-10; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Determine the maximum-tolerated dose (MTD) of BKM120 when administered orally in combination with daily bicalutamide and LH-RH agonists to men with non castrate metastatic prostate cancer | Patient follow-up done until progression, or until 6 months after the end of treatment

SECONDARY OUTCOMES:
Assess the efficacy of daily oral BKM120 in combination with LH-RH agonists and bicalutamide in men with NCMPC as measured by the overall rate and free survival of biological or clinical progression (composite measures). | Free survival of biological or clinical progression an expected average 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli Calmettes, Marseille, France

REFERENCES:
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr